CLINICAL TRIAL: NCT00905580
Title: Perioperative Administration of Pregabalin for Pain After Robot-assisted Endoscopic Thyroidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Severance Hospital, Anesthesia and Pain Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 4-2009-0070
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-10

CONDITIONS: Pain, Postoperative
Keywords: thyroidectomy; pain, postoperative; pregabalin
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients receive oral Placebo 150 mg 1 hour prior to surgery, and 12 hours later
  Interventions: Drug: Vitamin Complex (placebo)
- Pregabalin (Experimental): Patients receive oral pregabalin 150 mg 1 hour prior to surgery, and 12 hours later
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150 mg orally
  Arms: Pregabalin
Drug: Vitamin Complex (placebo) — Vitamin Complex 150 mg orally
  Arms: Placebo

SUMMARY:
The investigators hypothesize that pregabalin will decrease post-operative pain scores and analgesic use following robot-assisted endoscopic thyroidectomy compared to placebo. The primary outcome will be acute postoperative pain, measured by a verbal numerical rating score (VNRS) and total analgesic consumption during postoperative 48 hours. The secondary outcome will be the incidence of chronic pain and hypoesthesia in the anterior chest at 3 months after operation.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesia physical status class I & II
2. Age ≥ 20 and ≤ 65 years
3. Robot- assisted endoscopic thyroidectomy

Exclusion Criteria:

1. Known or suspected allergy, sensitivity, or contraindication to pregabalin or any of the standardized medications
2. Body mass index ≥ 40 kg/m2
3. History of seizure disorder
4. Current therapy with pregabalin, gabapentin, or any opioid
5. Any other physical or psychiatric condition which may impair their ability to cooperate with post-operative study data collection
6. Insulin-dependent diabetes mellitus
7. Renal insufficiency (estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim SY, Jeong JJ, Chung WY, Kim HJ, Nam KH, Shim YH. Perioperative administration of pregabalin for pain after robot-assisted endoscopic thyroidectomy: a randomized clinical trial. Surg Endosc. 2010 Nov;24(11):2776-81. doi: 10.1007/s00464-010-1045-7. Epub 2010 Apr 8. PMID 20376496

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients receive oral Placebo 1 hour prior to surgery, and 12 hours later
- Pregabalin: Patients receive oral pregabalin 1 hour prior to surgery, and 12 hours later
Period: Overall Study
Arm/Group | Placebo | Pregabalin
Started | 49 | 50
Completed | 47 | 47
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 50 | 99
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.5 (9.5) | 38.0 (8.2) | 38.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 48 | 94
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores (VNRS) at 1, 6, 24, 48 Hours Postoperatively.
Description: Pain was evaluated using an 11-point verbal numerical rating scale (VNRS). Patients were instructed preoperatively to express their pain on the 0-10 VNRS, where 0 means no pain at all, and 10 represents the worst pain imaginable
Time Frame: 1, 6, 24 & 48 hours
Measure: Median (Inter-Quartile Range); unit: VNRS
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 47 | 47
VNRS
  1 Hour | 6 [5 to 8] | 6 [4 to 8]
  6 Hour | 3 [2 to 4] | 2 [1 to 3]
  24 Hour | 2 [1 to 3] | 1 [1 to 2]
  48 Hour | 2 [1 to 2] | 1 [1 to 1]

2. Primary Outcome: The Number of Participants With the Indicated Side Effects - Nausea & Vomiting, Sedation, Headache, Dizziness Etc.
Description: Nausea and vomiting was graded on a four-point scale, where 0 = no nausea, 1 = mild nausea, 2 = severe nausea requiring antiemetics, and 3 = retching and/ or vomiting. Grades 3 and 4 were grouped together as postoperative nausea and vomiting (PONV) and rescue anti-emetic, metoclopramide 10 mg i.v. was given. We asked patients about sedation, headache, dizziness, blurred vision.
Time Frame: 1, 6, 24 & 48 hours
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 47 | 47
participants
  PONV | 10 | 7
  headache | 11 | 8
  dizziness | 6 | 14
  sedation | 1 | 6
  blurred vision | 0 | 3

3. Secondary Outcome: Number of Patients With Hypoesthesia in the Anterior Chest at 3 Months After Operation.
Description: we checked Hypoesthesia in the anterior chest at 3 months after operation by phone.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 47 | 47
participants | 13 | 10

4. Primary Outcome: Number of Patients Who Required Additional Analgesics During the First 48 Hours Postoperatively
Time Frame: 1, 6, 24 & 48 hours
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 47 | 47
participants
  0-1 hour | 31 | 26
  1-6 hour | 17 | 7
  6 - 24 hour | 15 | 2
  24 - 48 hour | 7 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 6/47 | 21/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Pregabalin (N=47)
Sedation (General disorders) | 1 (1) | 6 (6)
Dizziness (General disorders) | 6 (6) | 14 (14)
Blurred vision (General disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No